CLINICAL TRIAL: NCT02839421
Title: Efficacy of Moxifloxacin, Amoxicillin+Metronidazole for Aggressive Periodontitis Treatment
Brief Title: Efficacy of Three Antibiotic Protocols for Aggressive Periodontitis Treatment
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Facultad Nacional de Salud Publica (Other)
Responsible Party: Principal Investigator, Carlos Martin Ardila Medina, Titular Professor, Facultad Nacional de Salud Publica
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 003
Record Dates: First submitted 2016-05-31; First posted 2016-07-21 (Estimated); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Aggressive Periodontitis
MeSH Terms: conditions — Aggressive Periodontitis | interventions — Tooth Exfoliation; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Scaling and Root Planing plus moxifloxacin (Experimental): The interventions are Scaling and Root Planing (SRP) combined with systemically administered moxifloxacin (MOX) 400 mg, once daily for 7 days.The experimental treatment group consist of SRP combined with systemically administered MOX at the dosage of 400 mg once daily for 7 days.One-stage full-mouth SRP under local anesthesia will be performed (using manual instruments and ultrasonic debridement) in approximately 2 h and half by the same experienced clinician.The endpoint of SRP will be a tactile smooth root surface. The adjunctive agent will start at the SRP visit. Subjects in the MOX group will be extensively informed about the intake of the prescribed medication.
  Interventions: Drug: Scaling and Root Planing combined with moxifloxacin
- Scaling and Root Planing plus amox-metro (Active Comparator): The active comparator is Scaling and Root Planing (SRP) combined with systemically administered Amoxicillin (amox) + Metronidazole (metro) 500 mg tid each one for 7 days. The active comparator group consist of SRP combined with systemically administered Amoxicillin (amox) + Metronidazole (metro) 500 mg tid each one for 7 days.
  One-stage full-mouth SRP under local anesthesia will be performed (using manual instruments and ultrasonic debridement) in approximately 2 h and half by the same experienced clinician.The endpoint of SRP will be a tactile smooth root surface. The adjunctive agent will start at the SRP visit. Subjects in the amox-metro group will be extensively informed about the intake of the prescribed medication.
  Interventions: Drug: Scaling and Root Planing combined with moxifloxacin
- Scaling and Root Planing plus placebo (Placebo Comparator): Scaling and Root Planing (SRP) + placebo once daily for 7 days. The placebo comparator group consist of SRP combined with systemically administered placebo once daily for 7 days. One-stage full-mouth SRP under local anesthesia will be performed (using manual instruments and ultrasonic debridement) in approximately 2 h and half by the same experienced clinician.The endpoint of SRP will be a tactile smooth root surface. The placebo agent will start at the SRP visit. Subjects in the placebo group will be extensively informed about the intake of the prescribed medication.
  Interventions: Drug: Scaling and Root Planing combined with moxifloxacin

INTERVENTIONS:
Drug: Scaling and Root Planing combined with moxifloxacin — Scaling and Root Planing combined with systemically administered moxifloxacin (MOX) 400 mg, once daily for 7 days
  Other Names: periodontal scaling

SUMMARY:
The aim of the present study is to evaluate the clinical and microbiological efficacy of moxifloxacin or amoxicillin plus metronidazole in one-stage scaling and root planing in treating generalized aggressive periodontitis. Forty five subjects will be randomly allocated to 3 treatment groups. Subgingival plaque samples will be analysed for cultivable bacteria. The primary outcome variable to determine the superiority of one treatment over the others would be differences between groups for means CAL changes at 6 months post-treatment. Secondary outcome variables include differences between therapies for the mean changes in the mean levels of PD and the proportion of BOP.

ELIGIBILITY:
Inclusion Criteria:

* Subjects ≤30 years of age
* minimum of six permanent teeth, with at least one site each with probing depth (PD) and clinical attachment level (CAL) ≥5 mm and a minimum of six teeth other than first molars and incisors with at least one site each with PD and CAL ≥5 mm.

Exclusion Criteria:

* diabetes
* cardiovascular diseases
* immunological disorders or any other systemic disease that could alter the course of periodontal disease.
* Pregnant or nursing women
* smoking
* allergy to amoxicillin, metronidazole, fluoroquinolones or moxifloxacin
* consumption of systemic antimicrobials or anti-inflammatory drugs in the last 6 months
* periodontal therapy during the last 6 months

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2015-12; Primary Completion 2019-05-31 (Estimated); Study Completion 2019-05-31 (Estimated)

PRIMARY OUTCOMES:
clinical attachment level | 3 and 6 months
  It was defined that the primary outcome variable to determine the superiority of one treatment over the other would be differences between groups for means Clinical Attachment Level changes at 6 months post-treatment. This is a measure assessing change between two time points .

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Medellín, Antioquia, Colombia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hammami C, Nasri W. Antibiotics in the Treatment of Periodontitis: A Systematic Review of the Literature. Int J Dent. 2021 Nov 8;2021:6846074. doi: 10.1155/2021/6846074. eCollection 2021. PMID 34790237